CLINICAL TRIAL: NCT00349271
Title: Multicenter Randomized Study Of Cell Therapy In Cardiopathies - Chagas Cardiomyopathy
Brief Title: Cell Therapy in Chagas Cardiomyopathy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Change the sample size due to smaller variance than expected
Sponsor: Ministry of Health, Brazil (Other Government)
Collaborators: Financiadora de Estudos e Projetos (Other)
Responsible Party: Principal Investigator, Bernardo Rangel Tura, Professor, Ministry of Health, Brazil
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMRTCC-CHG
Record Dates: First submitted 2006-07-05; First posted 2006-07-06 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Chagas Cardiomyopathy
Keywords: Chagas Cardiomyopathy; Dilated Cardiomyopathy; stem cells; Therapeutics; Randomized Controlled Trials
MeSH Terms: conditions — Chagas Cardiomyopathy; Cardiomyopathy, Dilated | interventions — Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Stem Cell therapy (Experimental): Stem Cell therapy
  Interventions: Procedure: Stem cell; Drug: Filgrastime (G-CSF)
- Standart therapy (Active Comparator): Standart therapy
  Interventions: Drug: Standart therapy

INTERVENTIONS:
Procedure: Stem cell — Stem cell
  Arms: Stem Cell therapy
Drug: Filgrastime (G-CSF) — Filgrastime (G-CSF)
  Arms: Stem Cell therapy
Drug: Standart therapy — All drug with clinical evidence of benefical effect in Chagas disease
  Arms: Standart therapy

SUMMARY:
The purpose of this study is to determine effect of cell therapy in patients with severe dilated cardiomyopathy

DETAILED DESCRIPTION:
This protocol describes a double-blind placebo controlled randomized clinical trial to evaluate the efficacy of bone marrow derived stem cell implants in 300 bazillion patients with dilated cardiomyopathy and heart failure in class III or IV of the New York Heart Association.

The primary endpoint of this study is to evaluate the effect of the autologous bone marrow stem cell implant in the increase of the ejection fraction of the left ventricle in comparison with a control group, under optimized therapy for dilated cardiomyopathy. Secondary endpoints will evaluate the alteration in NYHA functional class, mortality rate, physical capacity (by ergoespirometry), life quality (Minnesota questionnaire) and pulmonary congestion in dilated cardiomyopathy patients the received the autologous bone-marrow stem cell implant.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of dilated cardiomyopathy according to WHO criteria
* Syndromic heart failure in functional class III or IV of the NYHA
* Enrollment and continuous follow-up in cardiac out-patient clinic
* Adequate medical therapy after optimization therapy
* Echocardiogram with an ejection fraction equal to or less than 35% by Simpson's rule

Exclusion Criteria:

* Valvular diseases, except functional mitral or tricuspid reflow
* Coronariography showing a significant lesion (obstruction of at least 50% of the lumen in the troncus or the main arteries - LAD, CX, RC) in one or more arteries
* Serologic diagnosis for Chagas disease or at least two of the following criteria: epidemiology, right bundle branch block, anterior hemi-block, apical aneurism
* Sustained ventricular tachycardia
* Abusive use of alcohol or illicit drugs
* Pregnancy
* Use of cardio toxic drugs
* Any co-morbidity with impact in life expectancy in 2 years
* Renal function compromised (creatinine above 2 mg/dl)
* Definitive implant of pace-makers, resynchronizers and CDIs
* Heart failure with symptoms initiating less than 1 year ago
* Active systemic arterial hypertension or history of hypertension

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2006-01; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
increase of the ejection fraction of the left ventricle | 1 year

SECONDARY OUTCOMES:
Death by any cause within 1 year of intervention | 1 year
Difference in life quality as estimated by Minnesota living with Heart Failure Questionnaire at six months and baseline | 1 year
Difference in NYHA functional class at six months and baseline | six months
Percent number of patients that reached an absolute increase of 5% in ejection fraction at six and twelve months | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo R Santos, MD,PhD, Principal Investigator — Centro de pesquisa Gonzalo Muniz; Gilson Feitosa, MD, Principal Investigator — Hospital Santa Isabel
Locations (1):
- INCL - National Institute of Cardiology Laranjeiras, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Ribeiro Dos Santos R, Rassi S, Feitosa G, Grecco OT, Rassi A Jr, da Cunha AB, de Carvalho VB, Guarita-Souza LC, de Oliveira W Jr, Tura BR, Soares MB, Campos de Carvalho AC; Chagas Arm of the MiHeart Study Investigators. Cell therapy in Chagas cardiomyopathy (Chagas arm of the multicenter randomized trial of cell therapy in cardiopathies study): a multicenter randomized trial. Circulation. 2012 May 22;125(20):2454-61. doi: 10.1161/CIRCULATIONAHA.111.067785. Epub 2012 Apr 20. PMID 22523306